## **Study Protocol**

Effectiveness of Intelligent Rehabilitation Robot

Training System Combined With Repetitive Facilitative

Exercise on Upper Limb Motor Function After Stroke: a

Randomized Control Trial

**Registration number: NCT06435624** 

Proposed date: June 15, 2024

| Study Start | June 15, 2024 | | |
|---|---|---|---|
| Primary Completion | August 31, 2024 | | |
| Study Completion | August 31, 2024 | | |
| Objective | To investigate the effectiveness of Intelligent robotic-assisted training (IRAT) combined with Repetitive facilitative exercise (RFE) on upper limb motor function in stroke patients | | |
| Design | Randomized controlled trial | | |
| Ethical Board | Medical Ethics Management Committee of Nanjing Mingzhou Rehabilitation<br>Hospital | | |
| Approval Number | NJKF202401001 | | |
| Location | Nanjing Mingzhou Rehabilitation Hospital, 102 Yaohua New Village, Qixia District, Nanjing, Jiangsu, China | | |
| Randomization | Closed envelope method | | |
| Masking | Single blind design (Outcomes assessor) | | |
| Arms | IRAT group | RFE group | CT group |
| Enrollment | 30 | 30 | 30 |
| Interventions | IRAT (30min) + RFE (30min) | RFE (60min) | CT (60min) |
| Outcome Measures | Fugl-Meyer assessment for upper extremity Active participation proportion Trajectory deviation Trajectory tracking error | | |
| Inclusion Criteria | Patients (18 to 74 years old) who suffered a first or Second unilateral stroke;<br>Chronic stroke (over 6 months from the onset);<br>Obvious upper limb movement disorders (FMA-UE scores from 25 to 42);<br>Ability to understand and follow simple directions | | |
| Exclusion Criteria | Pregnant or lactating; Upper extremity contracture, pain, or trauma; Perceptual, apraxic, or cognitive deficits that lead to inability to follow verbal instructions; Unable to maintain sitting posture; Cerebellar lesion; Clinically unstable medical disorders; Inability to provide informed consent | | |

Sample size calculation: G\*power 3.1.9.7 software was used to calculate the sample size. Using the FMA-UE scores from a pilot study, we calculated the effect size f to be 0.374. With an alpha level of 0.05 and a power of 0.80, the total sample size was calculated to be 72.

Statistical analysis method: SPSS 21.0 software was used to calculate the demographic and outcome measures. The Shapiro-Wilk test was used to assess the distribution of quantitative variables. Since all variables followed a normal distribution, a one-way analysis of variance was performed to compare the three groups. For post-hoc test, Bonferroni correction was applied when equal variances were assumed, and Tamhane's T2 was used when equal variances were not assumed. A paired samples t - test was used to compare data before and after the intervention. The chi-square test was

with p values <0.05 considered statistically significant.

used to compare qualitative variable. All significance tests were two-tailed,